CLINICAL TRIAL: NCT03701373
Title: Maintenance Treatment With S-1 Versus Observation After First-line Chemotherapy in Patients With Advanced Gastric Cancer: a Randomized Phase II Study
Brief Title: Maintenance Treatment With S-1 in Gastric Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ruihua Xu, Professor, Principal Investigator, President, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-1 maintenance study
Record Dates: First submitted 2018-10-02; First posted 2018-10-10 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Gastric Cancer Stage IV; Cancer of Stomach
Keywords: Advanced Gastric Cancer; Maintenance; S-1; First-line treatment
MeSH Terms: conditions — Stomach Neoplasms | interventions — Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S-1 maintenance group (Experimental): S-1 maintenance
  Interventions: Drug: S-1 maintenance
- Observation group (Other): Observation without anti-tumor treatment
  Interventions: Other: Observation

INTERVENTIONS:
Drug: S-1 maintenance — S-1 maintenance till disease progression or untolerable toxicities, in oral doses of 40 mg (BSA<1.25 m2), 50 mg (1.25≤BSA<1.50 m2) and 60 mg (BSA≥1.50 m2) b.i.d. on days 1-14 for each 21-day cycle.
  Other Names: S-1 monotherapy maintenance
  Arms: S-1 maintenance group
Other: Observation — Observation without anti-tumor treatment
  Other Names: Observation without anti-tumor treatment
  Arms: Observation group

SUMMARY:
Gastric cancer remains the third leading cause of cancer-related death worldwide and is especially frequent in East Asia. Fluoropyrimidines are the backbone of first-line chemotherapy for advanced gastric cancer (AGC), and S-1 provides new option with its simplicity and convenience.

5-Fluorouracil (5-FU) was the only efficacious treatment for AGC before the nineties of the 20th century, and afterwards with the discovery of chemotherapy such as cisplatin, oxaliplatin, S-1 and capecitabine, response rate as well as survival had been improved greatly.

Most of AGC will progress after first-line treatment; therefore, seeking an efficient and low toxic maintaining regimen to prolong progression-free survival (PFS) becomes a hot topic in oncologic field. Some clinical researches demonstrated maintenance treatment for advanced colorectal cancer (CRC) and lung cancer. The investigators had conducted a phase III clinical trial that demonstrated capecitabine maintenance versus observation prolonged PFS significantly after first-line chemotherapy with FOLFOX or XELOX regimens in advanced CRC. In AGC, several retrospective studies revealed patients receiving 5-FU/leucovorin(LV), capecitabine, or trastuzumab maintaining therapy experienced significantly longer PFS than that stopped chemotherapy after first-line chemotherapy. Some one-arm phase II clinical trials found 5-FU/LV, capecitabine, S-1, capecitabine plus bevacirumab, or capecitabine plus bevacirumab plus trastuzumab maintenance seemed to yield sound PFS and good tolerance. However, there were no randomized controlled clinical trials for maintenance treatment of these regimens in AGC, except that a phase II Chinese randomized controlled trial of Uracil and Tegafur (UFT) versus observation experienced early termination.

Above all, so far, there is no data to demonstrate that regular 2-6 months of chemotherapy followed by maintenance treatment could prolong PFS and OS for AGC. S-1 is effective for gastric cancer, and was approved as palliative treatment for advanced gastric cancer and adjuvant treatment; in addition, with its relative less frequency of side effects and convenient oral administration, S-1 as maintenance regimen could be prone to be accepted by patients. Therefore, the current study is designed to investigate that S-1 as maintenance treatment after first-line palliative chemotherapy could improve PFS and OS for patients with advanced gastric cancer through a perspective randomized clinical study.

DETAILED DESCRIPTION:
Patients with AGC who achieved objective response or stable disease after 2-6 months of first-line chemotherapy were randomly assigned to one of two groups, to receive either S-1 (40 mg for BSA<1.25 m2, 50 mg for 1.25≤BSA<1.50 m2 and 60 mg for BSA≥1.50 m2 b.i.d. on days 1-14, q3w) as maintenance therapy or observation. The treatment will continue until disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years
* Eastern Cooperative Oncology Group performance status (ECOG PS) 0-1
* At least one measurable lesion according to the Response Evaluation Criteria in Solid Tumor (RECIST version 1.0)
* Histologically confirmed gastric cancer with inoperable locally advanced or recurrent and/or metastatic disease, not amenable to curative therapy
* No previous chemotherapy for metastatic GC was allowed, the interval after the end of adjuvant/neoadjuvant chemotherapy beyond 6 months was allowable
* Life expectancy of at least 3 months
* Adequate hematologic, hepatic and renal function. Neutrophil count ≥ 1.5 × 109/L; platelet count ≥ 100 × 109/L; Serum bilirubin ≤ 1.5 × upper limit of normal (ULN), AST or ALT ≤ 2.5 × ULN (or ≤ 5 × ULN in patients with liver metastases), alkaline phosphatase ≤ 2.5 × ULN (or ≤ 5 × ULN in patients with liver metastases, or ≤ 10 × ULN in patients with bone but no liver metastases); serum creatinine ≤ 1.5 × ULN；and albumin ≥ 25 g/L
* Patients who achieved objective response or stable disease after 2-6 month first-line chemotherapy
* The first-line chemotherapy regimens were doublets including platinum (cisplatin or oxaliplatin) plus fluoropyrimidine (5-FU, capecitabine, or S-1)
* Signed informed consent

Exclusion Criteria:

* Known hypersensitivity to platinum (cisplatin or oxaliplatin) or fluoropyrimidine (5-FU, capecitabine, or S-1)
* History or clinical evidence of brain metastases
* Previous chemotherapy for metastatic disease
* Positive serum pregnancy test in women of childbearing potential
* Subjects with reproductive potential not willing to use an effective method of contraception
* Received any investigational drug treatment within 4 weeks of start of study treatment
* Other prior malignancies in the past 5 years
* Unresolved bowel obstruction or malabsorption syndrome

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
maintenance progression-free survival (PFS) | from date of randomization to maintenance or observation until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  The Kaplan-Meier survival from randomization to maintenance or observation until the date of first documented progression or date of death from any cause, whichever came first.

SECONDARY OUTCOMES:
progression-free survival from induction treatment (PFS2) | from induction treatment (the initiation date of first-line chemotherapy) until the date of first documented progression or date of death from any cause after maintenance treatment or observation, whichever came first, assessed up to 2 years
  The Kaplan-Meier survival from induction treatment (the initiation date of first-line chemotherapy) until the date of first documented progression or date of death from any cause after maintenance treatment or observation, whichever came first
overall survival (OS) | from induction treatment (the initiation date of first-line chemotherapy) until death from any cause or the last follow-up date, assessed up to 2 years.
  The Kaplan-Meier survival from induction treatment (the initiation date of first-line chemotherapy) until death from any cause or the last follow-up date.
toxicity relevant to S-1 maintenance/observation | from date of randomization to maintenance or observation until the date of first documented progression or unaccepted toxicities, assessed up to 30 days after the last oral administration of S-1.
  any toxicities occurring during the treatment of S-1 maintenance/observation

CONTACTS AND LOCATIONS:
Overall Officials: Rui-hua Xu, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li W, Zhao X, Wang H, Liu X, Zhao X, Huang M, Qiu L, Zhang W, Chen Z, Guo W, Li J, Zhu X. Maintenance treatment of Uracil and Tegafur (UFT) in responders following first-line fluorouracil-based chemotherapy in metastatic gastric cancer: a randomized phase II study. Oncotarget. 2017 Jun 6;8(23):37826-37834. doi: 10.18632/oncotarget.13922. PMID 27980221
- [Background] Qiu MZ, Wei XL, Zhang DS, Jin Y, Zhou YX, Wang DS, Ren C, Bai L, Luo HY, Wang ZQ, Wang FH, Li YH, Yang DJ, Xu RH. Efficacy and safety of capecitabine as maintenance treatment after first-line chemotherapy using oxaliplatin and capecitabine in advanced gastric adenocarcinoma patients: a prospective observation. Tumour Biol. 2014 May;35(5):4369-75. doi: 10.1007/s13277-013-1574-5. Epub 2014 Feb 11. PMID 24515655
- [Background] Petrioli R, Francini E, Roviello F, Marrelli D, Miano ST, Fiaschi AI, Laera L, Bellini MA, Roviello G. Treatment of advanced oesophagogastric cancer with FOLFOX-4 regimen followed by leucovorin/bolus and continuous infusion 5-FU as maintenance chemotherapy in patients aged >/= 75 years with impaired performance status. J Geriatr Oncol. 2015 Sep;6(5):380-6. doi: 10.1016/j.jgo.2015.06.002. Epub 2015 Jul 27. PMID 26228711
- [Background] Eren OO, Ozturk MA, Sonmez OU, Oyan B. Safety, Feasibility, and Efficacy of Capecitabine Maintenance in Patients With Advanced Gastric Cancer: A Retrospective Study. Am J Ther. 2016 Nov/Dec;23(6):e1493-e1497. doi: 10.1097/MJT.0000000000000156. PMID 25397587
- [Background] Chen J, Shen W, Xia J, Xu R, Zhu M, Xu M. [Effect of S-1 maintenance chemotherapy following DCF regimen in patients with advanced gastric cancer]. Nan Fang Yi Ke Da Xue Xue Bao. 2014 Jun;34(7):1057-60. Chinese. PMID 25057084
- [Background] Meulendijks D, de Groot JW, Los M, Boers JE, Beerepoot LV, Polee MB, Beeker A, Portielje JE, Goey SH, de Jong RS, Vanhoutvin SA, Kuiper M, Sikorska K, Pluim D, Beijnen JH, Schellens JH, Grootscholten C, Tesselaar ME, Cats A. Bevacizumab combined with docetaxel, oxaliplatin, and capecitabine, followed by maintenance with capecitabine and bevacizumab, as first-line treatment of patients with advanced HER2-negative gastric cancer: A multicenter phase 2 study. Cancer. 2016 May 1;122(9):1434-43. doi: 10.1002/cncr.29864. Epub 2016 Mar 11. PMID 26970343
- [Background] Meulendijks D, Beerepoot LV, Boot H, de Groot JW, Los M, Boers JE, Vanhoutvin SA, Polee MB, Beeker A, Portielje JE, de Jong RS, Goey SH, Kuiper M, Sikorska K, Beijnen JH, Tesselaar ME, Schellens JH, Cats A. Trastuzumab and bevacizumab combined with docetaxel, oxaliplatin and capecitabine as first-line treatment of advanced HER2-positive gastric cancer: a multicenter phase II study. Invest New Drugs. 2016 Feb;34(1):119-28. doi: 10.1007/s10637-015-0309-4. Epub 2015 Dec 8. PMID 26643663
- [Background] Palacio S, Loaiza-Bonilla A, Kittaneh M, Kyriakopoulos C, Ochoa RE, Escobar M, Arango B, Restrepo MH, Merchan JR, Rocha Lima CM, Hosein PJ. Successful use of Trastuzumab with anthracycline-based chemotherapy followed by trastuzumab maintenance in patients with advanced HER2-positive gastric cancer. Anticancer Res. 2014 Jan;34(1):301-6. PMID 24403478
- [Background] Luo HY, Li YH, Wang W, Wang ZQ, Yuan X, Ma D, Wang FH, Zhang DS, Lin DR, Lin YC, Jia J, Hu XH, Peng JW, Xu RH. Single-agent capecitabine as maintenance therapy after induction of XELOX (or FOLFOX) in first-line treatment of metastatic colorectal cancer: randomized clinical trial of efficacy and safety. Ann Oncol. 2016 Jun;27(6):1074-1081. doi: 10.1093/annonc/mdw101. Epub 2016 Mar 2. PMID 26940686